CLINICAL TRIAL: NCT00518102
Title: A Matched Cohort Study of Regranex (Becaplermin) and the Risk of Cancer
Brief Title: The Risk of Cancer in Users of Regranex (Becaplermin) and Matched Comparators (Nonusers of Regranex [Becaplermin])
Status: Completed | Type: Observational
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR012010; REGRANEX-EPI-01 (Other: Ethicon, Inc.)
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus
Keywords: REGRANEX (becaplermin); Platelet-derived growth factor BB; Cancer; Cancer incidence; Cancer mortality
MeSH Terms: conditions — Diabetes Mellitus; Neoplasms | interventions — Becaplermin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- 001: REGRANEX (becaplermin) A cohort of REGRANEX (becaplermin) users (ie patients treated with REGRANEX (becaplermin) a topical medication used to treat non-healing neuropathic foot ulcers in patients with diabetes).
  Interventions: Drug: REGRANEX (becaplermin)
- 002: REGRANEX (becaplermin) comparators A cohort of REGRANEX (becaplermin) nonusers (ie patients who are not treated with REGRANEX [becaplermin]) but are similar in characteristics to patients in the REGRANEX [becaplermin] user cohort)
  Interventions: Other: REGRANEX (becaplermin) comparators

INTERVENTIONS:
Drug: REGRANEX (becaplermin) — A cohort of REGRANEX (becaplermin) users (ie, patients treated with REGRANEX (becaplermin), a topical medication used to treat non-healing neuropathic foot ulcers in patients with diabetes).
  Groups: 001
Other: REGRANEX (becaplermin) comparators — A cohort of REGRANEX (becaplermin) nonusers (ie, patients who are not treated with REGRANEX [becaplermin]) but are similar in characteristics to patients in the REGRANEX [becaplermin] user cohort)
  Groups: 002

SUMMARY:
The purpose of this study is to compare the risk of cancers in patients who have used REGRANEX (becaplermin) to that of patients with similar characteristics and health issues who have not used REGRANEX (becaplermin). REGRANEX (becaplermin) is topical medication used to treat non-healing neuropathic foot ulcers in patients with diabetes.

DETAILED DESCRIPTION:
This is an observational retrospective study where data will be collected from a medical claims database derived from a large national managed care organization with over five million members. Members enrolled in a Medicare supplement program will also be included. The objective of this study is to determine the incidence of cancer among patients who have used REGRANEX (becaplermin) compared to patients who have not used REGRANEX (becaplermin). REGRANEX (becaplermin) is an FDA-approved prescription medicine that contains a platelet-derived growth factor that is used for the treatment of foot ulcers in patients with diabetes. Patients who were treated with REGRANEX (becaplermin) between January 1998 and June 2003 will be identified in a health insurance claims database. Another group of patients who have not been treated with REGRANEX (becaplermin) but have similar characteristics to patients treated with REGRANEX (becaplermin) will also be identified during the same time frame in the database. Medical record abstraction and review will be conducted to verify all incident cancers identified. Follow-up for study outcomes will be conducted from the date of accrual through termination of health-plan membership or December 2003 (whichever comes first). The date of accrual is the date of REGRANEX (becaplermin) exposure for each exposed patient and his or her matched unexposed comparison patients. Any incidence of death from cancer will also be identified. The primary outcome measure in the study will be the incidence rate of cancers of all kinds, grouped by organ site in patients who have used REGRANEX (becaplermin) and patients who have not used REGRANEX (becaplermin). A secondary objective is a similar comparison of the incidence of death from cancer. This is an observational study; no investigational drug will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Must have at least 6 months of continuous enrollment in health plan prior to Regranex initiation

Exclusion Criteria:

* Any cancer-related diagnoses identified in the claims data during baseline (the 6 month period prior to REGRANEX (becaplermin) initiation).

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with similar characteristics who were treated or who were not treated with REGRANEX (becaplermin) between January 1998 and June 2003 identified in a health insurance claims database.
Sampling Method: Probability Sample
Enrollment: 4431 (Actual)
Dates: Start 2003-01; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
The number of reported cases of cancers of all kinds, grouped by organ site in patients who have used REGRANEX (becaplermin) and patients who have not used not used REGRANEX (becaplermin). | From the date of accrual until the earliest of December 2003, outcome identification, health plan disenrollment, or death

SECONDARY OUTCOMES:
The number of reported deaths from cancer in patients who have used REGRANEX (becaplermin) and patients who have not used not used REGRANEX (becaplermin). | From the date of accrual until the earliest of December 2003, outcome identification, health plan disenrollment, or death

CONTACTS AND LOCATIONS:
Overall Officials: Ethicon, Inc. Clinical Trial, Study Director — Ethicon, Inc.

REFERENCES:
- See also: The Risk of Cancer in Users of REGRANEX (becaplermin) and Matched Comparators (Nonusers of REGRANEX [becaplermin]) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=217&filename=CR012010_REF.pdf